CLINICAL TRIAL: NCT00183391
Title: Measuring and Predicting Response to Atomoxetine and Methylphenidate
Brief Title: Stimulant Versus Nonstimulant Medication for Attention Deficit Hyperactivity Disorder in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jeffrey Newcorn, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 03-0612-00002; R01MH070935 (NIH); R01MH070564 (NIH); DSIR 84-CTM
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Child; Adolescent; School
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Atomoxetine (Active Comparator): Participants will receive treatment for ADHD with the non-stimulant atomoxetine
  Interventions: Drug: Atomoxetine; Drug: Methylphenidate
- Methylphenidate (Active Comparator): Participants will receive treatment for ADHD with the stimulant methylphenidate
  Interventions: Drug: Atomoxetine; Drug: Methylphenidate

INTERVENTIONS:
Drug: Atomoxetine — Participants will be randomly assigned to receive either methylphenidate or atomoxetine for either 2 or 5 weeks, depending on how soon they respond to the treatment. After the 2- or 5-week period, participants will be crossed-over to receive whichever medication they did not receive in the first part of the study.
Drug: Methylphenidate — Participants will be randomly assigned to receive either methylphenidate or atomoxetine for either 2 or 5 weeks, depending on how soon they respond to the treatment. After the 2- or 5-week period, participants will be crossed-over to receive whichever medication they did not receive in the first part of the study.

SUMMARY:
This study will determine the effectiveness of stimulant and nonstimulant medication in treating the symptoms of attention deficit hyperactivity disorder (ADHD) in children and adolescents.

DETAILED DESCRIPTION:
ADHD is one of the most frequently occurring disorders of children and adolescents and is a significant public health problem. The most common treatment for the condition is stimulant medication. However, there are an increasing number of children who are experiencing negative side effects from stimulants, such as dizziness, loss of appetite, and headaches; these side effects have made the need for alternative treatments all the more important. This study will compare the stimulant methylphenidate to the nonstimulant atomoxetine to determine which is more effective in treating ADHD symptoms in children and adolescents. The two medications differ in the neurotransmitters they influence. Stimulants such as methylphenidate act upon the neurotransmitter dopamine, while atomoxetine works on norepinephrine. It has been proposed that the difference in neurotransmitter stimulation may result in differences in an ADHD patient's response to treatment.

Participants will be randomly assigned to receive either methylphenidate or atomoxetine for between 4 to 6 weeks, depending on how soon they respond to the treatment. After the 4 to 6 week period, participants will be crossed-over to receive whichever medication they did not receive in the first part of the study.

Participants will have up to 14 weekly study visits. Over the first two visits, participants will undergo psychological and intelligence tests, a medical history, an electrocardiogram, blood and urine collection, and a physical exam. The remaining visits will occur weekly. During these visits, participants will receive their assigned medication and, along with their parents, will complete questionnaires about their response to treatment and any side effects they may be experiencing. The teachers of all participants will be asked to complete a questionnaire about their student's behavior at 4 different times during the study. Participant, parent, and teacher questionnaires will be used to assess the ADHD symptoms of participants, as well as self-report clinical scales completed by the participants.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV-TR criteria for ADHD
* Scores at least 1.5 standard deviation higher than age and gender mean on ADHD-RS keyed to ADHD subtype
* CGI Severity ADHD Rating greater than or equal to 4
* Currently attends school with at least 3 months left in high school
* Currently lives at home with parent(s) or legal guardian(s), now and for the past year before study entry, and is expected to remain there
* Normal physical exam, laboratory tests, and electrocardiogram
* Pulse and blood pressure within 95% of age and gender mean
* Full Scale IQ is greater than or equal to 75 OR if the results of testing indicate that Full Scale IQ is not a good indicator of intellectual ability, a General Ability Index greater than or equal to 75
* Weight is between 20 and 85 kilograms
* Able to swallow pills
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* History of atomoxetine or methylphenidate intolerance
* Any existing medical condition for which study medications are contraindicated
* If the child is in psychotherapy, no changes in therapy expected during the study trial
* Presence of any of the following: autism, mental retardation, schizophrenia, a psychotic disorder, bipolar disorder, severe depression, or conduct disorder
* Presence of a comorbid disorder that should be the primary focus of treatment
* Presence of a medical or neurological disorder precluding study medications or assessing ADHD
* Allergic reactions to multiple medications
* History of alcohol or drug abuse in the 3 months before study entry, or positive urine toxic screen that is not explained by a time limited medical circumstance
* Involved in a medication treatment study in the 30 days before study entry
* Female who is sexually active and is unwilling to use birth control
* Evidence of child abuse or neglect

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 232 (Actual)
Dates: Start 2005-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H. Newcorn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Mark A. Stein, PhD, Principal Investigator — University of Illinois, Chicago - Institute for Juvenile Research
Locations (2):
- United States (2):
  - University of Illinois, Chicago - Institute for Juvenile Research, Chicago, Illinois
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Result] Bedard AC, Stein MA, Halperin JM, Krone B, Rajwan E, Newcorn JH. Differential impact of methylphenidate and atomoxetine on sustained attention in youth with attention-deficit/hyperactivity disorder. J Child Psychol Psychiatry. 2015 Jan;56(1):40-8. doi: 10.1111/jcpp.12272. Epub 2014 Jun 19. PMID 24942409
- [Derived] Schulz KP, Bedard AV, Fan J, Hildebrandt TB, Stein MA, Ivanov I, Halperin JM, Newcorn JH. Striatal Activation Predicts Differential Therapeutic Responses to Methylphenidate and Atomoxetine. J Am Acad Child Adolesc Psychiatry. 2017 Jul;56(7):602-609.e2. doi: 10.1016/j.jaac.2017.04.005. Epub 2017 May 10. PMID 28647012

RESULTS

PARTICIPANT FLOW:
Groups:
- Atomoxetine Then Methylphenidate: Participants randomized to receive Atomoxetine until optimal response, then washed out and crossed-over to receive Methylphenidate.
- Methylphenidate Then Atomoxetine: Participants randomized to receive Methylphenidate until optimal response, then washed out and crossed-over to receive Atomoxetine.
Period: Block 1 - 5 Weeks
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Started | 108 | 124
Completed | 95 | 110
Not Completed | 13 | 14
Not completed — Withdrawal by Subject | 13 | 14
Period: Crossover Placebo - 2 Weeks
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Started | 95 | 110
Completed | 95 | 110
Not Completed | 0 | 0
Period: Block 2 - 5 Weeks
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Started | 95 | 110
Completed | 91 | 108
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine | Total
Number analyzed (Participants) | 108 | 124 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.34 (2.61) | 10.56 (2.83) | 10.41 (2.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 36 | 63
  Male | 81 | 88 | 169

OUTCOME MEASURES:

1. Primary Outcome: ADHD-RS Total Score
Description: ADHD-RS Total Score Attention Deficit Hyperactivity Disorder Rating Scale. Each item on the 18-item measure is scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms), yielding a possible total score of 0-54. Higher score indicates higher probability of diagnosis.
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Atomoxetine Then Methylphenidate: Block 1 receiving Atomoxetine first, washout period, then Block 2 receiving Methylphenidate
- Methylphenidate Then Atomoxetine: Block 1 receiving Methylphenidate first, washout period, then Block 2 receiving Atomoxetine
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
units on a scale
  Block 1 Baseline Week 0 | 39.58 (8.984) | 39.75 (9.835)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | 20.03 (13.657) | 17.59 (12.756)
  Block 2 Baseline Week 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline Week 8 | 34.32 (11.423) | 33.54 (12.077)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | 18.08 (12.192) | 22.13 (13.356)

2. Secondary Outcome: Treatment Preference Survey
Time Frame: Measured at ends of treatments one and two
Measure: Number; unit: percentage of participants
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
percentage of participants
  Treatment Preference of ATX | 41.8 | 27.4
  Treatment Preference of MPH | 50.5 | 51.9

3. Secondary Outcome: ADHD - H/I
Description: Attention deficit/hyperactivity disorder - hyperactivity/impulsivity (ADHD- H/I). Each item on the 18-item measure is scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms), yielding a possible total score of 0-27. Higher score indicates higher probability of diagnosis.
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
units on a scale
  Block 1 Baseline Week 0 | 16.56 (7.235) | 17.31 (7.887)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | 7.82 (7.159) | 7.24 (7.083)
  Block 2 Baseline 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline 8 | 13.99 (8.258) | 14.80 (8.310)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | 6.67 (5.818) | 8.87 (7.651)

4. Secondary Outcome: ADHD-RS Inattention
Description: Each item on the 18-item measure is scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms), yielding a possible total score of 0-27. Higher score indicates higher probability of diagnosis.
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
units on a scale
  Block 1 Baseline Week 0 | 23.30 (3.524) | 22.44 (4.027)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | 12.32 (7.889) | 10.35 (7.172)
  Block 2 Baseline Week 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline Week 8 | 20.33 (5.525) | 18.74 (5.572)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | 11.09 (7.103) | 13.26 (7.398)

5. Secondary Outcome: Clinical Global Impressions (CGI)- Severity
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
units on a scale
  Block 1 Baseline Week 0 | 5.14 (.756) | 5.09 (.716)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | 3.20 (1.641) | 2.83 (1.446)
  Block 2 Baseline Week 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline Week 8 | 4.75 (.938) | 4.55 (1.233)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | 2.94 (1.458) | 3.43 (1.460)

6. Secondary Outcome: Social Skills Rating Scale (SSRS)- Parent Version
Description: Measure of social skills, higher score is better. This scale is based on t-scores and does not have psychometrics available.
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
t-score
  Block 1 Baseline Week 0 | 82.71 (28.414) | 77.96 (22.779)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | 91.07 (35.350) | 88.57 (26.099)
  Block 2 Baseline Week 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline Week 8 | 78.58 (21.112) | 82.35 (28.698)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | 91.07 (33.887) | 87.96 (19.501)

7. Secondary Outcome: Child Conflict Index (CCI)
Description: Measure of conflict within the home over the past 24 hours. The CCI is a validated measure of family conflicts in the home and is completed by parents. It consists of 42 items (for boys) or 36 items (for girls) reflecting attention-seeking and conflictual behavior, as well as negativity and withdrawal. Items are scored as yes (1 point) or no (0 points). Mean score between 0 and 1 reported, with higher score indicating greater conflict.
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
units on a scale
  Block 1 Baseline Week 0 | .3224 (.19841) | .3385 (.19795)
  Block 1 End of Treatment week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment week 6 | .2386 (.21233) | .1978 (.20251)
  Block 1 End of Treatment Week 8: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 8 | .3526 (.20878) | .3078 (.20744)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | .2118 (.20053) | .2304 (.18978)

8. Secondary Outcome: Continuous Performance Test (CPT)
Description: CPT Commissions, impulsive responses, higher score is worse. This scale is based on t-scores and does not have psychometrics available.
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
T-scores
  Block 1 Baseline Week 0 | 51.3277 (9.73401) | 52.8976 (9.36961)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | 51.7005 (9.57790) | 51.1713 (9.96929)
  Block 2 Baseline Week 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline Week 8 | 59.8788 (8.82849) | 51.2159 (9.00827)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | 50.0763 (11.16765) | 49.1616 (10.02259)

9. Secondary Outcome: Children's Sleep Questionnaire
Description: Children's Sleep Problems Severity, sum of scores, higher is worse.The scale assessed contains 16 items, each scored 0 to 3, with 0 representing no problems and 3 representing daily problems. total range from 0 to 48. This score does not have psychometrics available.
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
units on a scale
  Block 1 Baseline Week 0 | 5.14 (.756) | 5.09 (.716)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | 3.20 (1.641) | 2.83 (1.446)
  Block 2 Baseline Week 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline Week 8 | 4.75 (.938) | 4.55 (1.233)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | 2.94 (1.458) | 3.43 (1.460)

10. Secondary Outcome: Assessment of Affective Range (AAR)
Description: Affective problems. This scale consists of 8 items, scored 0-3, with 0 representing no problems and 3 representing extreme problems. This analysis presents sum of scores, higher is worse. Full range from 0 to 24. This score does not have psychometrics available.
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
units on a scale
  Block 1 Baseline Week 0 | 11.2609 (2.85251) | 10.6905 (3.44309)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | 10.6889 (2.83495) | 10.8257 (2.77170)
  Block 2 Baseline Week 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline Week 8 | 9.7108 (2.99402) | 10.1400 (3.06831)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | 10.9886 (2.69736) | 10.9286 (3.02652)

11. Secondary Outcome: Tics: Total Motor
Description: Modified Yale Global Tic Severity Scale, sum, higher is worse. This score does not have psychometrics available. The Yale Global Tic Severity Scale (YGTSS) is a semistructured clinician-rated instrument that assesses the severity and frequency of motor and phonic tics over the previous week. Five index scores are obtained during the assessment, where higher scores indicate greater frequency or severity. These indices are: Total Motor Tic Score (0-25), Total Phonic Tic Score (0-25), Total Tic Score (0-50) Overall Impairment Rating (0-50).
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
units on a scale
  Block 1 Baseline Week 0 | .196 (.7727) | .111 (.4297)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | .053 (.2941) | 1.342 (11.3544)
  Block 2 Baseline Week 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline Week 8 | .000 (.0000) | .214 (.8494)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | .160 (.7656) | .143 (.6686)

12. Secondary Outcome: Tics: Total Phonic
Description: as for outcome 11
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
units on a scale
  Block 1 Baseline Week 0 | .161 (.5649) | .028 (.1655)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | .018 (.1325) | 1.329 (11.3542)
  Block 2 Baseline Week 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline Week 8 | .039 (.1960) | .057 (.2892)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | .060 (.3136) | .016 (.1260)

13. Secondary Outcome: Tics: Total Impairment
Description: as for outcome 11
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
units on a scale
  Block 1 Baseline Week 0 | 5.304 (22.4936) | .292 (1.8571)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | 1.737 (13.1129) | .132 (1.1471)
  Block 2 Baseline Week 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline Week 8 | .000 (.0000) | .643 (3.1762)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | .500 (2.9014) | .397 (2.2543)

14. Secondary Outcome: Vital Signs - Systolic Blood Pressure
Description: Systolic blood pressure - the amount of pressure in arteries during contraction of the heart muscle Normal range varies by age, sex, height and weight and can range from 80mm Hg to 130mmHg
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: mm HG
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
mm HG
  Block 1 Baseline Week 0 | 101.11 (11.877) | 101.60 (11.261)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | 102.10 (12.442) | 103.29 (12.374)
  Block 2 Baseline Week 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline Week 8 | 99.74 (12.199) | 101.29 (12.629)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | 102.34 (11.797) | 102.51 (11.488)

15. Secondary Outcome: Vital Signs - Diastolic Blood Pressure
Description: Diastole blood pressure - blood pressure when the heart muscle is between beats. normal range varies by age, sex, height and weight and can range from 34mm Hg to 90mmHg
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: mm HG
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
mm HG
  Block 1 Baseline Week 0 | 61.78 (8.773) | 61.26 (7.882)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | 64.58 (8.638) | 62.77 (8.609)
  Block 2 Baseline Week 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline Week 8 | 62.33 (7.835) | 61.28 (8.442)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | 62.82 (7.325) | 65.44 (8.699)

16. Secondary Outcome: Vital Signs - Pulse
Description: Heartbeats per minute. Range varies from 50-205 depending on age and level of activity.
Time Frame: up to 14 weeks
Population: see participant flow section for participants that did not complete blocks
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 108 | 124
beats per minute
  Block 1 Baseline Week 0 | 78.20 (12.927) | 77.49 (12.365)
  Block 1 End of Treatment Week 6: number analyzed (Participants) | 95 | 110
  Block 1 End of Treatment Week 6 | 84.46 (14.697) | 82.05 (12.915)
  Block 2 Baseline Week 8: number analyzed (Participants) | 95 | 110
  Block 2 Baseline Week 8 | 82.96 (13.931) | 81.30 (12.683)
  Blocks 2 End of Treatment Week 14: number analyzed (Participants) | 91 | 108
  Blocks 2 End of Treatment Week 14 | 84.85 (13.314) | 84.31 (13.095)

17. Secondary Outcome: SES (Hollingshead)
Description: Measure of socioeconomic status, score calculated from averaging likert responses, lower = worse
Time Frame: up to 14 weeks
Population: data not collected
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Conners-Wells Adolescent Self Report
Description: Standardized measure of ADHD symptoms and severity, norm referenced T scores, higher = worse
Time Frame: up to 14 weeks
Population: data not collected
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Conners Teacher Rating Scale- Short
Description: Standardized measure of ADHD symptoms and severity, norm referenced T scores, higher = worse
Time Frame: up to 14 weeks
Population: data not collected
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Child Behavior Checklist (CBCL)
Description: CBCL Total Score, measure of psychosocial problems, higher is worse.
Time Frame: Measured at screening
Population: data not collected
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Social Skills Rating Scale (SSRS)- Teacher Version
Description: as for outcome 6
Time Frame: up to 14 weeks
Population: data not collected
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Permanent Mathematics Product Test (PERMP)
Description: Measure of fluency in performance of simple mathematics, sum, lower = worse
Time Frame: up to 14 weeks
Population: data not collected
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Actigraphy
Description: Measure of physical activity
Time Frame: Measured daily throughout the study
Population: data not collected
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Sleep Logs
Description: Questionnaire, qualitative
Time Frame: Measured daily throughout the study
Population: data not collected
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Hyperactivity, Attention, and Learning Problems (HALP) Medical and Developmental History Questionnaire
Description: Questionnaire, qualitative designed to collect family history, prenatal environmental influences, and developmental history.
Time Frame: Measured at screening
Population: data not collected
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: HALP Rebound Effects Questionnaire
Description: Questionnaire, qualitative assesses symptoms of rebound (moodiness, irritability, aggression, and ADHD symptoms) when the medication wears off at night.
Time Frame: up to 14 weeks
Population: data not collected
Arm/Group | Atomoxetine Then Methylphenidate | Methylphenidate Then Atomoxetine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Block 1 ATX: Block 1 first four weeks received Atomoxetine
- Block 1 MPH: Block 1 first four weeks received Methylphenidate
- Block 2 ATX: Block 2 (weeks 8 to 13) received Atomoxetine
- Block 2 MPH: Block 2 (weeks 8 to 13) received Methylphenidate
Arm/Group | Block 1 ATX | Block 1 MPH | Block 2 ATX | Block 2 MPH
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/124 | 0/95 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/124 | 0/95 | 0/110
Other Adverse Events (participants affected / at risk) | 24/108 | 35/124 | 20/95 | 25/110
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Block 1 ATX (N=108) | Block 1 MPH (N=124) | Block 2 ATX (N=95) | Block 2 MPH (N=110)
Insomnia (General disorders) | 5 | 16 | 3 | 14
Aggression (Psychiatric disorders) | 6 | 6 | 5 | 4
Appetite Loss (Gastrointestinal disorders) | 7 | 9 | 7 | 4
Irritability (Psychiatric disorders) | 6 | 4 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No